CLINICAL TRIAL: NCT06381349
Title: Predicting Outcomes of Gastric Peroral Endoscopic Myotomy Using a Gastric Electrical Mapping System: GPOEM-GEMS
Brief Title: Predicting Outcomes of GPOEM Using Gastric Electrical Mapping
Acronym: GPOEM-GEMS
Status: Recruiting | Type: Observational
Sponsor: Chris Varghese (Other)
Responsible Party: Sponsor-Investigator, Chris Varghese, Lead Clinical Investigator, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Other Study IDs: GPOEM-GEMS
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-05

CONDITIONS: Gastroparesis
Keywords: endoscopy; electrophysiology; phenotyping
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult patients with gastroparesis: 1. Provision of signed and dated informed consent form understand the risks and benefits of the study
  2. Aged ≥18 years old
  3. Patients must be clinically selected for GPOEM at their respective study site.
  4. Patients are undergoing their index GPOEM procedure
  Interventions: Diagnostic Test: Gastric Alimetry test

INTERVENTIONS:
Diagnostic Test: Gastric Alimetry test — Gastric Alimetry test will be performed within 30-days prior to G-POEM procedure. It's results will not inform clinical management in this observational study.

SUMMARY:
Gastric peroral endoscopic myotomy (GPOEM) is a minimally-invasive procedure that involves dividing the pylorus, to enhance gastric emptying in gastroparesis patients. This is a single-arm, multi-centre, prospective observational study to determine the clinical utility of Gastric Alimetry in predicting GPOEM treatment outcomes. The investigators further aim to develop a clinical decision rule to inform patient selection. Gastric Alimetry will be conducted <1 month prior to GPOEM. All subjects will then be followed up for 12 months.

DETAILED DESCRIPTION:
This protocol proposes no change to the clinical management of patients which is left to the discretion of the patients' primary clinical team.

Patients as part of this study will undergo a baseline assessment via Gastric Alimetry, and concurrent symptom, quality of life, and health psychology questions.

GPOEM will be performed as per standard site protocol, with data captured in RDCap.

Patients will be followed up at 1-month, 3-month, 6-months, and 12-months using the myCap (REDCap) app.

Participants and clinicians can opt-in for a repeat Gastric Alimetry test at 6 or 12 months following their GPOEM procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Indicated for GPOEM

Exclusion Criteria:

* Pregnant or breast-feeding
* Inability to perform Gastric Alimetry test: history of severe skin allergies or sensitivity to cosmetics or lotions; chronically damaged or vulnerable epigastric skin (fragile skin, wounds, inflammation); patients unable to remain in a relaxed reclined position for the test duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-years or older with gastroparesis awaiting a G-POEM procedure that are able to undergo Gastric Alimetry testing.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom Index (GCSI) | 6 months
  ≥ 1 decrease in total GCSI score [higher score = worse symptoms]

SECONDARY OUTCOMES:
Patient Assessment of Upper GastroIntestinal Disorders-Quality of Life (PAGI-QoL) | 1, 3, 6, and 12 months
  0 - 5; higher score = better quality of life
EQ-5D scores | 1, 3, 6, and 12 months
  0 - 1; higher score being better quality of life
Patient assessment of upper gastrointestinal disorders-symptom severity index (PAGI-SYM) | 1, 3, 6, and 12 months
  0 - 1; higher score being increased symptom burden
Patient Health Questionnaire - 8 (PHQ-8) | 6, and 12 months
  0 - 12; higher score being increased depression severity
Generalized Anxiety Disorder 7-item (GAD-7) | 6, and 12 months
  0 - 21; higher score indicates increased anxiety
Perceived Stress Scale 4 (PSS-4) | 6, and 12 months
  0 - 16; higher scores indicate higher stress
Brief Illness Perception Questionnaire-Revised | 6, and 12 months
  0 - 80; higher scores indicate worse illness perception
Alimetry® Gut-Brain Wellbeing (AGBW) | 1, 3, 6, and 12 months
  0 - 40; higher scores indicate higher mental health burden
Work Productivity and Activity Impairment (WPAI) | 12 months
  0-100%; higher scores indicating increased loss of work productivity and activity impairment

OTHER OUTCOMES:
Change in Gastric Alimetry Phenotype | 6
  Change in phenotype classification on repeat Gastric Alimetry testing before and after G-POEM

CONTACTS AND LOCATIONS:
Locations (1):
- University of Auckland, Auckland, Auckland, New Zealand